CLINICAL TRIAL: NCT00051909
Title: Efficacy and Safety of LY451395 in Patients With Probable Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6764; H6N-MC-LEAM
Record Dates: First submitted 2003-01-17; First posted 2003-01-20 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — N-((2-(4'-(2-(methylsulfonyl)amino)ethyl)(1,1'-biphenyl)-4-yl)propyl)-2-propanesulfonamide

INTERVENTIONS:
Drug: LY451395

SUMMARY:
Study of an investigational medication for the treatment of Alzheimer's Disease in patients who are not taking Aricept, Reminyl, Exelon.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical diagnosis of Alzheimer's Disease
* Must be at least 50 years of age
* Must fluently read and speak English
* Must have a reliable caregiver

Exclusion Criteria:

* Has serious health problems other than Alzheimer's Disease
* Cannot swallow whole pills
* Has had a menstrual period in the last two years
* Takes insulin for diabetes
* Has taken Aricept, Reminyl, or Exelon in the last 5 weeks

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-11; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Beverly Hills, California
  - Fresno, California
  - Boca Raton, Florida
  - Fort Lauderdale, Florida
  - Miami Beach, Florida
  - Boston, Massachusetts
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Wichita Falls, Texas